CLINICAL TRIAL: NCT05380596
Title: Impact of TelePharmaceutical Care on People With Type 2 Diabetes Melitus, Seen at the Special Medicines Pharmacy of the State of Rio Grande do Sul: a Randomized Clinical Trial (TelePharmaceutical Care Diabetes Trial)
Brief Title: TelePharmaceutical Care Diabetes Trial
Acronym: TPCDT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rio Grande do Sul State Health Department - SES/RS (Other Government)
Collaborators: Agnes Nogueira Gossenheimer (Unknown); Ana Paula Rigo (Unknown); Roberto Eduardo Schneiders (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RioGrandeSulSHD
Record Dates: First submitted 2022-05-09; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Diabete Mellitus; Diabete Type 2; Telemedicine; Telehealth
Keywords: Telehealth; Pharmaceutical care; Diabetes mellitus; Pharmaceutical services; Tele-interventions
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This is an unblinded randomized clinical trial comparing the outcomes between a group that will receive a Pharmaceutical Telecare intervention (pharmaceutical consultation via telephone), and the control group that will receive only the usual care. All steps of this study will follow the recommendations of the CONSORT guideline for clinical trials (SCHULZ, 2010)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (No Intervention): Patients in the control group will remain out of contact with the research group and will receive usual care, which consists of receiving medications without additional information. After completion of the project, the control group will receive educational materials related to the care of people with diabetes and, if the effectiveness of the Pharmaceutical Telecare service is proven, this possibility of care will be offered to users.
- Intervention (Active Comparator): The intervention will be carried out through three teleconsultations, one per month, with a pharmacist (Times 0, 1, 2 and 3), via cell phone. Each consultation will address an aspect of health education for DM2.
  Interventions: Behavioral: Telepharmaceutical Care

INTERVENTIONS:
Behavioral: Telepharmaceutical Care — The intervention will be carried out through three teleconsultations, one per month, with a pharmacist (Times 0, 1, 2 and 3). In the opportunities, aspects related to pharmacotherapy and health status, non-pharmacological approaches, treatment adherence and evaluation of problems related to pharmacotherapy (PRM) will be discussed.
  Arms: Intervention

SUMMARY:
The prevalence of Diabetes Mellitus (DM) in the world is currently around 9.3% of adults aged between 20 and 79 years, which corresponds to 463 million people living with DM, and about 80% of these people are found in developing countries. In Brazil, fourth in the number of patients with Type 2 Diabetes Mellitus (DM2) in the world, the prevalence of DM is around 12%, with a significant increase in the last three decades. Non-adherence to DM treatment is known as a problem in the scenario and internationally, as it impairs the physiological response to the disease, increasing the direct and indirect cost of treatment. Pharmaceutical care is a practice model characterized by the provision of pharmaceutical services that optimize treatment, improve the process of medicines used, and aim at their best use. With the calamity situation arising from the COVID-19 pandemic created in the state of Rio Grande do Sul, the Pharmaceutical Telecare service was implemented. Dapagliflozin was recently incorporated into the Brazilian public system for the treatment of type 2 DM. Considering that there are no studies in Brazil to date on the use, treatment adherence, and problems related to pharmacotherapy (PRM) associated with dapagliflozin, and also considering that the guidance and monitoring of patients remotely have become more frequent and necessary, the purpose of this protocol is to describe a clinical trial that will evaluate the impact of a pharmaceutical telecare service in aspects related to treatment adherence, disease control, and costs, offered to people with DM2 using dapagliflozin. The hypothesis that will be tested is that Pharmaceutical Telecare can be as effective as standard care for type 2 diabetes and assess the associated costs related to teleconsultation in public health settings.

ELIGIBILITY:
Inclusion Criteria:

* People aged 18 years or older, with a previous diagnosis of type 2 diabetes mellitus and who take dapagliflozin at the Special Medicines Pharmacy of the State of Rio Grande do Sul, Brazil, will be selected. In addition, it will be considered an inclusion criterion that the person is available to receive phone calls.

Exclusion Criteria:

* Do not present a telephone record registered in the system;
* Be participating in another diabetes education program;
* Pregnancy;
* Severe cognitive problems;
* Communication difficulties;
* Presence of other injuries;
* Patients who are hospitalized at the time of recruitment will also be excluded from participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Variation in HbA1c levels | 3 months
  The patient'S blood glucose level
Adherence to treatment - Brief Medication Questionnaire (BMQ) | 3 months
  Assessment of treatment adherence through the BMQ.

SECONDARY OUTCOMES:
Adherence to treatment | 3 months
  Assessed by the Self-Care Inventory - revised (SCI-R).
Variation in blood pressure levels | 3 months
  Will be obtained from medical records and laboratory tests that patients report at the beginning of tele calls.
Variation in lipid profile | 3 months
  Will be obtained from medical records and laboratory tests that patients report at the beginning of tele calls.
Hospitalizations | 3 months
  Number of hospitalizations in the period.
Medical consultations | 3 months
  Number of medical consultations performed.
Emergency visits | 3 months
  Number of emergency visits.
Drug-related problems | 3 months
  Number of drug-related problems found and resolved.
Service-related cost | 3 months
  Service-related cost
Quality of life measured by DQOL-Brazil; | 3 months
  Quality of life measured by Diabetes Quality of Life Measure (DQOL-Brasil).

CONTACTS AND LOCATIONS:
Locations (1):
- Rio Grande do Sul State Health Department - SES/RS, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No